CLINICAL TRIAL: NCT01336790
Title: The International Lymphatic Disease and Lymphedema Patient Registry and Biorepository
Brief Title: International Lymphatic Disease and Lymphedema Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: Lymphatic Education & Research Network (Unknown)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Other Study IDs: SU-04052011-7662; 16384 (Other: Stanford IRB)
Record Dates: First submitted 2011-04-07; First posted 2011-04-18 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lymphedema
Keywords: Lymphatic disease; Lymphedema; Lymphangiomatosis; Lymphangiectasia; Protein-losing enteropathy; Vascular Anomalies
MeSH Terms: conditions — Lymphedema; Lymphatic Diseases; Lymphangiectasis; Protein-Losing Enteropathies; Vascular Malformations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the International Lymphatic Disease and Lymphedema Patient Registry and Biorepository is to collect health information in order to study the disease classification, natural history, and impact of Lymphatic Disease, Lymphedema and Related Disorders and its treatments and medical outcomes.

DETAILED DESCRIPTION:
This project represents the inauguration of an International Patient Registry for Lymphatic Diseases. This project will be completed through an affiliation with the Lymphatic Education & Research Network, a non-profit organization whose mission is to promote research and the development of new therapies for patients with lymphatic diseases, including lymphedema. The registry will provide researchers with much-needed clinical data to study the impact of diseases of the lymphatic system, in order to develop improved treatments and find a cure for lymphatic diseases, lymphedema, and related disorders. The establishment of this initiative is a major step forward in research for direct study of groups of patients with lymphatic disease. In the future, this project will be able to be linked with a biorepository, in which tissue and blood samples derived from patients will be made available for research into human disease states. An international patient registry and tissue/cell bank program paves the way for future clinical trials of experimental drugs and therapies designed to treat lymphatic disease in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lymphatic disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants (national and international participants) with the presence of lymphatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-03; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of lymphatic disease | 15 years

SECONDARY OUTCOMES:
socioeconomic impact of lymphatic disease | 15 years
  The data in the registry will be utilized to determine the financial impact of requisite diagnostic and treatment interventions and will be analyzed to consider the relative contribution of third-party payer participation in the cost of care. The financial impact of disease and treatment will be addressed through the financial data entered by registry participants.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
grouped data may be shared

REFERENCES:
- See also: The International Lymphatic Disease Patient Registry will serve as a repository of information that will enhance the future ability of health care professionals to accurately identify, categorize, treat and prevent lymphatic disease. — https://lernregistry.stanford.edu/